CLINICAL TRIAL: NCT05089578
Title: Examination of the Use of Integrative Treatment Methods by Individuals Undergoing COVID-19 Acording to the Health Promotion Model: a Sample Qualitative Study
Brief Title: Integrative Treatment Methods in COVID-19
Status: Completed | Type: Observational
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, nurhandogan, Asisst.Prof., Amasya University
Other Study IDs: Amasya U-2
Record Dates: First submitted 2021-10-20; First posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: COVID-19; Patient Experience; Health Attitude
Keywords: Covid-19; patient experince; integrative treatment; qualitative study; health promotion model
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Individuals with Covid-19: Interviews were conducted with individuals who had Covid-19, and their experiences with the integrative methods they used were determined.
  Interventions: Other: focus interview

INTERVENTIONS:
Other: focus interview — The "Information Form" including descriptive characteristics of the individuals undergoing Covid-19, the semi-structured "Interview Form", and the Complementary Therapy Use Form were used as the data collection tools. The Information Form consisted of 13 questions including socio-demographic and disease-related characteristics of individuals. In-depth interview method was used to collect data. Interviews were held by organizing video calls and online meeting programs on mobile phones both due to pandemic measures and in order to enable individuals to communicate comfortably. The time period in which the individuals felt most ready for the interview was determined and the data were collected during that time. During the interview, effective communication techniques were used, active listening was carried out and individuals were guided using question forms in accordance with the aim of the study. The interviews lasted for an average of 25-30 minutes.

SUMMARY:
This study was conducted to examine the use of integrative treatment methods by individuals undergoing Covid-19. In this study, which was designed in the qualitative and phenomenological type, the criterion sampling method was used and 12 people were included in the sample.

DETAILED DESCRIPTION:
This study was a qualitative type of phenomenological study conducted to examine the use of integrative treatment methods by individuals undergoing Covid-19. The study was completed with 12 people. The data were collected between July and October 2021. The interviews lasted for an average of 25-30 minutes. The data collected with the semi-structured interview form were analyzed by descriptive content analysis method after the interviews were over.

ELIGIBILITY:
Inclusion Criteria:

* individuals who underwent Covid-19 and used any of the integrative treatment methods
* agreed to participate in the study constituted the sample group.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who underwent Covid-19 and used any of the integrative treatment methods constituted the population of the study. Using the criterion sampling method, individuals who underwent Covid-19 and used any of the integrative treatment methods and agreed to participate in the study constituted the sample group. In accordance with the nature of qualitative research, the study was completed with 12 people.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Using integrative treatment method | 15 July- October 2021
  All participants included in the study had used at least one of the integrative treatment methods.
Kind of integrative treatment methods | October 2021
  It was determined that vitamin C and medicinal plants were frequently used in addition to their medical treatments.

CONTACTS AND LOCATIONS:
Overall Officials: Gamze Fıskın, PhD, Principal Investigator — Amasya University; Nurhan Dogan, PhD, Principal Investigator — Amasya University
Locations (1):
- Amasya University Sciences Faculty, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No